CLINICAL TRIAL: NCT06225115
Title: A First in Human Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of KYN-5356 in Adult, Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of KYN-5356 in Healthy Subjects Aged 18 to 55 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kynexis B.V. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYN5356-CL-001
Record Dates: First submitted 2023-12-20; First posted 2024-01-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Dysfunction; Schizophrenia
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- SAD Cohort 1 (Experimental): Single-Ascending Dose Cohort 1. Intervention: KYN-5356 A mg or placebo, single dose, oral tablet
  Interventions: Drug: KYN-5356; Drug: placebo
- SAD Cohort 2 (Experimental): Single-Ascending Dose Cohort 2. Intervention: KYN-5356 B mg or placebo, single dose, oral tablet
  Interventions: Drug: KYN-5356; Drug: placebo
- SAD Cohort 3 (Experimental): Single-Ascending Dose Cohort 3. Intervention: KYN-5356 C mg or placebo, single dose, oral tablet
  Interventions: Drug: KYN-5356; Drug: placebo
- SAD Cohort 4 (Experimental): Single-Ascending Dose Cohort 4. Intervention: KYN-5356 D mg or placebo, single dose, oral tablet
  Interventions: Drug: KYN-5356; Drug: placebo
- SAD Cohort 5 (Experimental): Single-Ascending Dose Cohort 5. Intervention: KYN-5356 E mg or placebo, single dose, oral tablet
  Interventions: Drug: KYN-5356; Drug: placebo
- MAD Cohort 1 (Experimental): Multiple-Ascending Dose Cohort 1. Intervention: KYN-5356 G mg or placebo, oral tablets for 7 days
  Interventions: Drug: KYN-5356; Drug: placebo
- MAD Cohort 2 (Experimental): Multiple-Ascending Dose Cohort 2. Intervention: KYN-5356 H mg or placebo, oral tablets for 7 days
  Interventions: Drug: KYN-5356; Drug: placebo
- MAD Cohort 3 (Experimental): Multiple-Ascending Dose Cohort 3. Intervention: KYN-5356 I mg or placebo, oral tablets for 7 days
  Interventions: Drug: KYN-5356; Drug: placebo
- Food Effect Cohort (Experimental): Intervention: KYN-5356 J mg, single dose, oral tablets in fasted or fed state.
  Interventions: Drug: KYN-5356

INTERVENTIONS:
Drug: KYN-5356 — KYN-5356, oral tablet
Drug: placebo — placebo, oral tablet
  Arms: MAD Cohort 1; MAD Cohort 2; MAD Cohort 3; SAD Cohort 1; SAD Cohort 2; SAD Cohort 3; SAD Cohort 4; SAD Cohort 5

SUMMARY:
This first-in-human clinical trial with a randomized, double-blind, placebo-controlled, dose-escalation study design is regarded as standard to test the safety, tolerability, and pharmacokinetics of KYN-5356.

The study comprises 3 parts:

Part 1: Single Ascending Dose study Part 2: Multiple Ascending Dose study Part 3: Food Effect study

The aim of Parts 1 and 2 of the study is to evaluate the safety and tolerability following single and multiple ascending doses of KYN-5356.

The secondary aim is to evaluate the pharmacokinetics (PK) of escalating single and multiple doses of KYN-5356. In Part 2, cerebrospinal fluid will be sampled to explore PK and pharmacodynamic effects of KYN-5356.

The potential effect of food intake on the disposition of KYN-5356 following a single oral dose will be evaluated in Part 3. Part 3 is an open-label, randomized, 2 period, 2 sequence design.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study procedures and agrees to participate by providing written informed consent prior to any study procedures.
* Subject is between 18 and 55 years of age (inclusive), on the date of signing the informed consent form.
* Subject has a body mass index between 18 and 30 kg/m2, inclusive.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential or a woman of childbearing potential who agrees to follow the contraceptive guidance (highly effective birth control method) from Screening until end of the study. Note: Males should use appropriate contraceptive method from Screening until end of the study.
* Subject is judged to be in good health by the Principal Investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory safety tests.
* Subject is willing to adhere to the study requirements and restrictions.

Exclusion Criteria:

* Subject has positive serology for HBsAg, HCV, or HIV, or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the Investigational Medicinal Product.
* Subject has any illness judged by the Principal Investigator as clinically significant, in the 3 months prior to first dosing of the Investigational Medicinal Product.
* Subject has a suicidality score of "yes" on item 4 or item 5 of the suicidal ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the suicidal behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the suicidal behavior section), if this behavior occurred in the past 2 years.
* Subject has a history or current sign or symptom of psychiatric or neurologic disease.
* Subject has a history of head trauma in the past year and/or current seizures.
* Subject is a smoker (use of tobacco products in the previous 3 months from Screening) or uses nicotine or nicotine-containing products and has a positive urine cotinine test at Screening or Admission.
* Subject has a history of alcohol and/or illicit drug abuse within 2 years of entry or has a positive screening test for alcohol and/or drugs of abuse at Screening or Admission.
* Subject consumes caffeine containing beverages exceeding 500 mg caffeine per day (5 cups of coffee) during the off-site days during the study.
* Subject has regular excessive consumption of alcohol within 6 months prior to Screening (7 drinks/week for females, 14 drinks/week for males where 1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor).
* Subject has a history or current sign or symptom of a cardiovascular, renal, or metabolic bone disease or disease of bone remodeling, or any history of endocrine disease, including an abnormal laboratory result for pre-specified clinical laboratory safety parameters related to these conditions.
* Subject has a history or presence of clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction. A first-degree atrioventricular block will not be considered as a significant abnormality. Subject has QTcF > 450 ms (mean values per parameter will be considered) detected on the 12-lead ECG at Screening or Admission.
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance <85 mL/min, using the Cockcroft-Gault formula), or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs at Screening or Admission.
* Subject has a history of malignancy within the past 5 years prior to Screening with the exception of excised and curatively treated non-metastatic cell carcinoma of the skin which is considered cured with minimal risk of recurrence.
* Subject tests positive for SARS-CoV-2 at Admission.
* Additional exclusion criteria for subjects in the MAD Part in view of lumbar puncture for cerebrospinal fluid (CSF) sampling and the ERP assessment.
* Subject uses any prescription drugs, herbal supplements, within 4 weeks prior to initial dosing, and/or over-the-counter medication, dietary supplements (vitamins included) within 2 weeks prior to initial dosing, other than what is allowed per protocol.
* Subject received vaccination 1 month before admission or plans to receive vaccination during the study.
* Use of other investigational drugs/devices within 5 half-lives of the drug from enrollment (time of the subject signing the informed consent form), or within 30 days, whichever is longer.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to initial dosing.
* Plasma donation (> 200 mL) within 7 days prior to first dosing.
* Resting vital signs at Screening (blood pressure > 140/90 mmHg, heart rate > 90 beats per minute, respiratory rate > 20 breaths per minute, and clinically significant elevated body temperature), or any clinically significant abnormalities in vital signs requiring intervention in the opinion of the Investigator. Up to 2 repeat measurements are permitted to confirm eligibility.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | Initiation of dosing through the last follow-up visit after the last dose, approximately 8 days in the MAD and 5 days after dosing in the SAD and the Food Effect parts of the study
  All cohorts

SECONDARY OUTCOMES:
PK parameters: Cmax [SAD] | Baseline (predose) through 72 hours post dosing
  Maximum plasma concentration determined directly from the concentration-time profile. For each dose in SAD part.
PK parameters: tmax [SAD] | Baseline (predose) through 72 hours post dosing
  Time of maximum plasma concentration determined directly from the concentration-time profile. For each dose in SAD part.
PK parameters: AUCinf [SAD] | Baseline (predose) through 72 hours post dosing
  Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time calculated using the linear-log trapezoidal rule. For each dose in SAD part.
PK parameters: Cmax on Day 1 [MAD] | Baseline (predose) through 24 hours post first dosing
  Maximum plasma concentration determined directly from the concentration-time profile. For each dose in MAD part
PK parameters: tmax on Day 1 [MAD] | Baseline (predose) through 24 hours post first dosing
  Time of maximum plasma concentration determined directly from the concentration-time profile. For each dose in MAD part.
PK parameters: Cmax,ss [MAD] | Baseline (predose) through 96 hours post dosing on Day 7.
  Maximum observed plasma concentration during a dosing interval at steady state. For each dose in MAD part.
PK parameters: tmax,ss [MAD] | Baseline (predose) through 96 hours post dosing on Day 7.
  Time of maximum plasma concentration determined directly from the concentration-time profile at steady state. For each dose in MAD part.
PK parameters: AUCtau on Days 1 and 7 [MAD] | Baseline (predose) through 96 hours post dosing on Day 7.
  Area under the concentration-time curve over the dosing interval. For each dose in MAD part
PK parameters: AUCinf [MAD] | Baseline (predose) through 96 hours post dosing on Day 7.
  Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time calculated using the linear-log trapezoidal rule. For each dose in MAD part.

CONTACTS AND LOCATIONS:
Overall Officials: Hakop Gevorkyan, MD, MBA, Principal Investigator — Parexel
Locations (1):
- Parexel Los Angeles Early Phase Clinical Unit, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No